CLINICAL TRIAL: NCT02781259
Title: Selective Lymph Node Dissection Using Fluorescent Dye in Node-positive Breast Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Seok Won Kim, Associate professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-01-046-007
Record Dates: First submitted 2016-05-08; First posted 2016-05-24 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Breast Neoplasms
Keywords: Sentinel Lymph Node Biopsy; Fluorescence; Breast Neoplasms; Indocyanine Green
MeSH Terms: conditions — Breast Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Selective Lymph Node Dissection (Experimental): 10cc of 20μg/mL indocyanine green is injected at the nipple-areola complex before surgery. Routine axillary lymph node dissection is performed. Acquired lymph nodes are separated to fluorescent positive lymph nodes and fluorescent negative lymph nodes with imaging devices.
  Interventions: Procedure: Axillary lymph node dissection; Drug: Indocyanine green; Device: Imaging devices

INTERVENTIONS:
Procedure: Axillary lymph node dissection — Lymph node dissection is performed in axillary lymph node level I and II. In case of palpable nodes in level II, additional lymph node dissection in level III is done.
Drug: Indocyanine green — 10cc of 20μg/mL indocyanine green is injected at the nipple-areola complex before surgery
  Other Names: Diagnogreen
Device: Imaging devices — Near-infrared fluorescence is collected by imaging lenses and digital camera.

SUMMARY:
In this study, navigation of lymphatic passage after sentinel lymph node with indocyanine green was performed during axillary lymph node dissection in breast surgery . By comparing the concordance between the passage of indocyanine green and actual lymph node metastasis, selective lymph node dissection can be developed.

DETAILED DESCRIPTION:
Low dose of indocyanine green emits near-infrared fluorescence, which can penetrate thin tissues like breast or skin. The operator can track the lymphatic pathway without skin incision in real time. By these characteristics, indocyanine green is currently used for sentinel lymph node biopsy in breast cancer surgery. Indocyanine green can also stain lymph nodes beyond the sentinel lymph nodes. This is why we can identify the lymphatic metastasis pathway of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Operable breast cancer patient
* Preoperatively axillary lymph node positive proven patients or sentinel lymph node positive patients whom requires axillary lymph node dissection

Exclusion Criteria:

* Breast cancer history
* Occult breast cancer
* Past history of axillary surgery
* Iodine hypersensitivity
* Pregnancy

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-02 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Number of metastatic lymph nodes in fluorescent positive lymph nodes and fluorescent negative lymph nodes confirmed by pathologist | within 2 weeks (plus or minus 3 days) after surgery
  Concordance analysis is done by comparing lymph node metastasis between fluorescent positive lymph nodes and fluorescent negative lymph nodes.

SECONDARY OUTCOMES:
Clinicopathological factors associated with lymph node metastasis in fluorescent negative lymph nodes | within 2 weeks (plus or minus 3 days) after surgery
  Risk factor analysis of fluorescent negative lymph node with positive lymph node metastasis

CONTACTS AND LOCATIONS:
Overall Officials: SeokWon Kim, MD. PhD., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung medical center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No